CLINICAL TRIAL: NCT03218553
Title: Effects of Perioperative Administration of Dexamethasone on Postoperative Complications and Mortality After Non-cardiac Major Surgery : a Randomized, Multicentre, Double Blind, Study
Brief Title: Effects of Perioperative Administration of Dexamethasone on Postoperative Complications and Mortality After Non-cardiac Major Surgery
Acronym: PACMAN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RC17_0029
Record Dates: First submitted 2017-07-10; First posted 2017-07-14 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Major Non-cardiac Surgery
MeSH Terms: interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexamethasone (Experimental): Standard cares plus postoperative administrations of glucocorticoid
  Interventions: Drug: Dexamethasone
- placebo (Placebo Comparator): Standard cares plus postoperative administrations of placebo
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Dexamethasone — Dexamethasone : first dose : 0,2mg.kg-1 at the end of the surgical procedure, second dose (0,2 mg.kg-1) 24 hours after the surgery
  Arms: Dexamethasone
Drug: Placebos — placebo : first infusion at the end of the surgical procedure, second 24 hours after the surgery
  Arms: placebo

SUMMARY:
Postoperative complications are major healthcare problems and are associated with a reduced short-term and long-term survival after surgery. Major surgery is associated with a predictable and usually transient Systemic Inflammatory Response (SIRS), depending on the magnitude of the surgical trauma. An excessive SIRS syndrome participates to the development of postoperative organ dysfunction, infection and mortality. Corticosteroids may decrease the postsurgical SIRS in cardiac surgery: in a large multicenter randomized trial, a single intravenous administration of high-dose dexamethasone did not reduce the incidence of a composite endpoint of adverse events but was associated with a reduced incidence of postoperative pulmonary complications and infections and with a reduction in hospital stay. However, a similar study, recently published in the Lancet was negative. Evidences from one meta-analysis, including 11 studies of moderate quality (439 patients in total), suggest that intraoperative administration of corticosteroids during major abdominal surgery decreases postoperative complications, including infectious complications, without significant risk of anastomotic leakage. At present, no large randomized controlled trial has been performed in patients undergoing major non-cardiac surgery. In acute medicine, several lines of evidence have shown that low to moderate doses of corticosteroids decrease the excessive inflammatory response, without inducing immuno suppression. However, despite the widespread use of corticosteroids to reduce postoperative nausea and vomiting and to improve analgesia, concerns continue to be raised about their safety, especially regarding an increased risk of postoperative infection.

We hypothesize that the perioperative administration of glucocorticoids would reduce postoperative morbidity after major non-cardiac surgery through dampening of the inflammatory response. Given the number of surgical patients for whom the question applies, the study is of significant clinical importance

DETAILED DESCRIPTION:
Background :

Postoperative complications are major healthcare problems and are associated with a reduced short-term and long-term survival after surgery. Corticosteroids may decrease the postsurgical SIRS in cardiac surgery, but this treatment is not recommended yet. The aim of the current study is to assess the efficiency and the safety of dexamethasone to prevent on postoperative complications.

Methods :

The PACMAN trial is a multicenter, randomized, controlled, double-blind, two-arms study. 1222 patients undergoing major surgery (duration >90 minutes and one or more risk factor of postoperative complication) are randomized to dexamethasone (0.2mg/kg at the end of the surgery and at day1) or to placebo. The primary outcome is a composite outcome of major postoperative complication during 14 days after the surgery.

Analyzes will be conducted, first, on data from the intention-to-treat (ITT) population, second, in the modified intention-to-treat (mITT) population as well as in the per-protocol population. All statistical analyzes will take into account stratified randomization (cancer and type of surgery) and will be adjusted on the center as random effect as.

Discussion :

The PACMAN trial is the first randomized controlled trial powered to investigate whether perioperative administration of dexamethasone in high risk patients improve outcomes.

ELIGIBILITY:
Inclusion Criteria:

Major surgery (> 90 minutes and realized under general anesthesia) of the abdomen, pelvis, thorax, face/neck, vascular surgery in a patient older than 65 years Or Major surgery (> 90 minutes and realized under general anesthesia) of the abdomen, pelvis, thorax, face/neck, vascular surgery in a patient older than 50 years and presenting one of the following criteria

* Presence of a defined risk factor for cardiac or respiratory disease (exercise tolerance equivalent to 6 metabolic equivalents or less)
* Medical history of stroke
* Moderate to severe renal impairment (clearance of creatinine ≤ 30 mll/L)
* Active smoking
* Averaged observed blood losses over 500 ml
* Emergency surgery

Exclusion Criteria:

* Pregnant women, Minors, Adults under guardianship or trusteeship
* Treatment with systemic corticosteroids at a dose > 5 mg.day-1 of equivalent prednisolone in the previous 3 months
* Patients with chronic renal failure (clearance of creatinine < 10 ml/min)
* Patients for which death is deemed imminent and inevitable or patients with an underlying disease process with a life expectancy of less than 1 month
* Patient with preoperative shock (defined by the need for vasoactive drugs before surgery)
* Acute Pulmonary edema in the last 7 days
* Active bacterial or viral infection
* Allergy to the intravenous formulation of dexamethasone
* Uncontrolled psychotic disorder (acute or chronical)

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1222 (Actual)
Dates: Start 2017-12-13 (Actual); Primary Completion 2019-04-16 (Actual); Study Completion 2019-04-16 (Actual)

PRIMARY OUTCOMES:
Composite outcome at least one item among the following:-Postoperative sepsis, severe sepsis, septic shock-Postoperative pulmonary complication: pneumonia, need for invasive and/or noninvasive ventilation for respiratory failure-All-cause mortality | 14 days

SECONDARY OUTCOMES:
All cause mortality | 28 days
Hospital free days | 28 days
Rate of patients with post operative sepsis | 28 days
Postoperative intubation rate for respiratory failure | 28 days
  Postoperative respiratory failure requiring invasive ventilation
Rate of patients with postoperative respiratory failure requiring non-invasive ventilation | 28 days
Surgical complications | 28 days
  The Clavien-Dindo classification
Duration of hospitalization | 28 days
Rate of unplanned hospitalization in intensive care unit | 28 days
Rate of patients developing postoperative organ failures | 28 days
Blood level of marker of inflammation (C Reactive protein) | 28 days
Delayed healing defined as non hermetic scar | 28 days
ICU length of stay | 28 days
Rate of patients with Gastric ulcer | 28 days
Rate of patients with Digestive bleeding | 28 days
Rate of patients with Anastomotic leakage | 28 days
Dose of insulin | 3 days
Rate of patients with Hypokaliemia (< 4 mmol/l) | 28 days
Rate of patients with Dysnatremia (<139 mmol/l or > 145 mmol/l) | 28 days
Rate of patients with Hypocalcemia (<2.2 mmol/l) | 28 days
Rate of patients with Cardiac events (Atrial fibrillation / cardiac flutter, Acute coronary syndrome or Cardiac failure) | 28 days

CONTACTS AND LOCATIONS:
Locations (29):
- France (29):
  - CHU Angers, Angers
  - CHU La Cavale Blanche, Brest
  - Hôpital Estaing, CHU de Clermont Ferrand, Clermont-Ferrand
  - Hôpital Beaujon, Clichy
  - CHD Vendée, La Roche-sur-Yon
  - Centre Hospitalier Du Mans, Le Mans
  - Hôpital Claude Huriez, Lille
  - Hopital Edouard Herriot, Lyon
  - Institut Paoli Calmettes, Marseille
  - Hôpital Timone, Marseille
  - Hôpital Nord, Marseille
  - Hôpital Saint-Eloi, Montpellier
  - Clinique Jules Verne, Nantes
  - Le Confluent, Nantes
  - Hotel Dieu Nantes, Nantes
  - Hôpital Laennec, Nantes
  - C.R.L.C.C. Nantes Atlantique, Nantes
  - Hôpital Saint Antoine, Paris
  - Hôpitaux Universitaires Saint-Louis, Lariboisière, Fernand Widal, Paris
  - CHU Lyon Sud, Pierre-Bénite
  - CHU de Poitiers, Poitiers
  - Ch Quimper, Quimper
  - Hôpital Pontchaillou, Rennes
  - CHU de Rouen, Rouen
  - CHU Saint Etienne, Saint-Etienne
  - Nouvel Hôpital Civil, Strasbourg
  - CHU de Toulouse, Toulouse
  - CH Valenciennes, Valenciennes
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Asehnoune K, Le Moal C, Lebuffe G, Le Penndu M, Josse NC, Boisson M, Lescot T, Faucher M, Jaber S, Godet T, Leone M, Motamed C, David JS, Cinotti R, El Amine Y, Liutkus D, Garot M, Marc A, Le Corre A, Thomasseau A, Jobert A, Flet L, Feuillet F, Pere M, Futier E, Roquilly A; PACMAN study group. Effect of dexamethasone on complications or all cause mortality after major non-cardiac surgery: multicentre, double blind, randomised controlled trial. BMJ. 2021 Jun 2;373:n1162. doi: 10.1136/bmj.n1162. PMID 34078591
- [Derived] Asehnoune K, Futier E, Feuillet F, Roquilly A; PACMAN group. PACMAN trial protocol, Perioperative Administration of Corticotherapy on Morbidity and mortality After Non-cardiac major surgery: a randomised, multicentre, double-blind, superiority study. BMJ Open. 2019 Mar 23;9(3):e021262. doi: 10.1136/bmjopen-2017-021262. PMID 30904834